CLINICAL TRIAL: NCT05153096
Title: A Phase I, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of NBL-015 in Patients With Advanced Solid Tumors
Brief Title: Evaluation of the Safety and Efficacy of NBL-015 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NovaRock Biotherapeutics, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBL-015-CSP-001
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: solid tumors (Experimental): Dose-escalation stage: Patients will receive NBL-015 once every two or three weeks, starting at a dose of 1 mg/kg.
  Cohort-expansion stage: Patients will receive NBL-015 at selected dose as per the results of dose-escalation stage.
  Interventions: Drug: NBL-015

INTERVENTIONS:
Drug: NBL-015 — NBL-015 by intravenous infusion

SUMMARY:
This trial is an open-label, multicenter, dose-escalation and cohort-expansion Phase I clinical study in patients with advanced solid tumors. The aim of this study is to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of NBL-015 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a multicenter, open-label phase I clinical trial conducted in patients with CLDN18.2-positive advanced solid tumors, aiming to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of NBL-015 in patient with advanced solid tumors.

This study consists of two stages: the stage I (dose escalation and dose expansion) and the stage II (NBL-015 monotherapy cohort expansion and combination of NBL-015 with standard treatment cohort expansion).

The dose escalation phase is divided into 5 dose levels. NBL-015 is escalated in order of 1 mg/kg, 3 mg/kg, 10 mg/kg, 20 mg/kg, 30 mg/kg until MTD. If MTD is still not observed in the preset highest dose group, the investigator and the sponsor can jointly decide whether to conduct a higher dose group study. If necessary, intermediate doses may be conducted. The first dose group (1 mg/kg) is the accelerated titration group, in which 1 patient will be enrolled, and the "3+3" dose escalation design will be followed from the second dose group.

If RP2D can be determined based on clinical study data in the dose escalation stage, Stage II cohort expansion will be directly conducted. Alternatively, based on the safety, tolerability and efficacy data obtained from dose-escalation studies, dose expansion and different dosing can be explored if necessary.

Based on available PK and clinical efficacy data, appropriate dose groups will be selected for cohort expansion. The cohort expansion stage includes the NBL-015 monotherapy cohort expansion trial and the combination of NBL-015with standard treatment cohort expansion trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤75 years, (subject to the date of signing the informed consent) who voluntarily sign the informed consent.
2. Positive expression of Claudin 18.2 which is defined as moderate to severe membrane staining (2+/3+) in ≥50% of tumor cells tested by central laboratory immunohistochemistry (IHC).
3. Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors.
4. At least one measurable lesion as per RECIST version 1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
6. Life expectancy ≥12 weeks.
7. Adequate major organ function within 7 days prior to treatment.
8. Serum pregnancy tests were negative in women of reproductive age (WOCBP) within 7 days prior to initial use of the investigational drug. Patients and their spouses must agree to take adequate contraceptive measures from the time of signing the informed consent until 6 months after the last dose. During this period, women are not breastfeeding and men avoid sperm donation.

Exclusion Criteria:

1. A history of other malignancies within 3 years prior to first dose, except for locally curable cancers.
2. Patients with central nervous system metastases.
3. Gastrointestinal abnormalities include:

   A) Pyloric obstruction or persistent recurrent vomiting (defined as ≥3 times of vomiting in 24 hours); B) There is a high risk of gastrointestinal bleeding or that there are other gastrointestinal abnormalities affecting the drug toxicity assessment determined by the investigator.
4. Patient with a history of serious cardiovascular disease.
5. A history of severe autoimmune disease that the investigator judged inappropriate for inclusion.
6. Patients with active hepatitis B or C, or active syphilis infection, or HIV positive.
7. Patients who are known to have severe allergic reactions and/or contraindications to prescription ingredients of NPL-015 or monoclonal antibodies, or who are intolerant to combination drugs;
8. Patients who underwent major surgery (excluding needle biopsy) within 4 weeks prior to initial use of the investigational drug, or who required elective surgery during the trial period, or who had severe unhealed wounds, traumatic ulcers, etc.
9. Toxicity of previous antitumor therapy did not return to grade 1 or below (CTCAE V5.0), except for toxicity of alopecia and other toxicity that researchers judged to have no safety risk.
10. Patients have previously been treated with a drug targeting Claudin18.2.
11. The time interval between the last anti-tumor treatment and the first use of experimental drug should meet the following requirements:

    A) Received antitumor therapy such as chemotherapy, radiotherapy (except local radiation therapy for pain relief), targeted therapy, immunotherapy, and other investigational agents within 4 weeks prior to initial administration; B) Received oral fluorouracil, small-molecule targeted drugs and traditional Chinese medicine with anti-tumor indications within 2 weeks prior to initial administration.
12. Receiving a corticosteroid (prednisone>10 mg/ day or equivalent dose of the same kind of drug) or other immunosuppressant treatment, except for:

    A) Local, ocular, intraarticular, intranasal, and inhaled glucocorticoids; B) Short-term use of glucocorticoids for prophylactic treatment (e.g. to prevent contrast allergy).
13. Live attenuated vaccine is received within 2 weeks prior to the first use of the investigational drug or is planned for the study period.
14. Other conditions that the investigator considers inappropriate for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Approximately 4 years
  Incidence of adverse events (AEs) of single and multiple dose (according to NCI CTCAE 5.0).An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Incidence of serious adverse events (SAEs) | Approximately 4 years
  Incidence of serious adverse events (SAEs) of single and multiple dose (according to NCI CTCAE 5.0).
Maximum tolerated dose (MTD) (if available) | Approximately 1 year
  MTD is defined as the prior dose level below the dose level at which 2/6 subjects suffer dose limiting toxicities.
Dose Limiting Toxicity (DLT ) | Up to 28 days after first injection
  Dose-limiting toxicity in patients with advanced tumors treated by NBL-015.
Recommended Phase 2 dose (RP2D) | Approximately 2 years
  RP2D will be determined using available safety and efficacy data.
Objective response rate (ORR) (in stage Ⅱ) | Approximately 2 years in stage Ⅱ
  Percentage of participants with CR or PR.
Disease control rate (DCR) (in stage Ⅱ) | Approximately 2 years in stage Ⅱ
  Percentage of participants with CR or PR or SD.
Duration of response (DOR) (in stage Ⅱ) | Approximately 2 years in stage Ⅱ
  DOR is defined as the time from first objective response (CR or PR per RECIST v 1.1) to first occurrence of objective tumor progression (progressive disease per RECIST v 1.1) or death from any cause, whichever occurs first.
Progression-free survival (PFS) (in stage Ⅱ) | Approximately 2 years in stage Ⅱ
  PFS is defined as the time from first dose to the first observation of disease progression (based on central reading) or death from any cause (as assessed by the independent reviewer).
Overall survival (OS) (in stage Ⅱ) | Approximately 2 years in stage Ⅱ
  OS is defined as the time from first dose to death from any cause.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Maximum plasma drug concentration (Cmax)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Area under the concentration time curve from 0 to time t (AUC0-t)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Area under the concentration time curve from 0 to the last measurable point (AUClast)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Area under the concentration time curve from 0 to infinity (AUC0-inf)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Time to maximum concentration (Tmax)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Elimination half-life (t1/2)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Volume of Distribution During the Terminal Phase (Vz)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Clearance (CL)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Terminal elimination rate constant (λz)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Mean residence time in the body from 0 to the time t of the last quantifiable drug concentration (MRT0-t)
Pharmacokinetic (PK) | Up to 21 Days after the sixth injection in stage I, after the fifth injection in stage II.
  Mean Residence time from 0 to infinite (MRT0-Inf)
Incidence of anti-drug antibody (ADA) | Once before each of the first five doses and once every 3 months thereafter, and 30 Days after the last dose.
  Number of positive participants with ADA positive.
Objective response rate (ORR) (in stage Ⅰ) | Approximately 2 years in stage Ⅰ
  Percentage of participants with CR or PR.
Disease control rate (DCR)(in stage Ⅰ) | Approximately 2 years in stage Ⅰ
  Percentage of participants with CR or PR or SD.
Duration of response (DOR)(in stage Ⅰ) | Approximately 2 years in stage Ⅰ
  DOR is defined as the time from first objective response (CR or PR per RECIST v 1.1) to first occurrence of objective tumor progression (progressive disease per RECIST v 1.1) or death from any cause, whichever occurs first.
Progression-free survival (PFS) (in stage Ⅰ) | Approximately 2 years in stage Ⅰ
  PFS is defined as the time from first dose to the first observation of disease progression (based on central reading) or death from any cause (as assessed by the independent reviewer).
Overall survival (OS) (in stage Ⅰ) | Approximately 2 years in stage Ⅰ
  OS is defined as the time from first dose to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided